CLINICAL TRIAL: NCT01211561
Title: Colon Cancer Prevention Using Selenium
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Dr. Richard Benya, University of Illinois
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 2008-1122
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2010-09-29 (Estimated); Status verified 2010-09

CONDITIONS: Prevention of Colorectal Cancer
MeSH Terms: interventions — Selenium; Selenomethionine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Selenium, selenomethionine (Experimental)
  Interventions: Drug: Selenium, selenomethionine
- placebo (Active Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Selenium, selenomethionine — Patients will receive one 200 ug pill of Selenomethionine
  Arms: Selenium, selenomethionine
Drug: placebo — Patients will be given one 200 ug placebo pill each day for 6 months
  Arms: placebo

SUMMARY:
Selenium's ability to prevent colorectal cancer (CRC) has been suspected for nearly 30 years, but has never been directly studied in humans. The investigators will directly assess selenium's ability to prevent CRC by measuring alterations in aberrant crypt foci (ACF), an accepted surrogate marker for CRC.

ACF's are very small (i.e., microscopic) collections of abnormally shaped cells that are a commonly used marker of CRC risk. Screening colonoscopy at UIC routinely uses methods that allow ACF counting to be done as a part of standard practice. ACF's are not fixed, like polyps or cancers, but can disappear as a person's risk for developing CRC decreases.

The investigators propose giving patient's with 6 or more ACF's 200 mcg selenized yeast or placebo, and determining if there is a drug-dependant decrease in ACF number. The primary objective is to determine whether selenized yeast supplementation, compared to placebo, causes significant reduction of ACF number from baseline levels. The primary endpoint will be change in ACF number

ELIGIBILITY:
Inclusion Criteria:

- All non-pregnant patients >50 years of age

Exclusion Criteria:

* The following will be specifically looked for, and result in patients not being eligible for study enrollment:

  * Use of non-steroidal anti-inflammatory drugs or glucocorticosteroids within 60 days of study entry.
  * History of chronic IBD or prior pelvic radiation (inflammation distorts crypt pattern).
  * Intake of any selenium supplements within 60 days of study entry, including vitamins.
  * Patients with increased bleeding risk from biopsy protocol (i.e. renal failure, decompensated cirrhosis, blood dyscrasia).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in ACF biomarkers | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard V Benya, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago Medical Center, Chicago, Illinois, United States